CLINICAL TRIAL: NCT01559714
Title: BE STRONG HCM: Biomarkers, Exercise Stress Testing, and mRi to Obtain New insiGhts in Hypertrophic CardioMyopathy Study
Brief Title: A Biomarker and MRI Study on Troponin Release After Exercise in Hypertrophic Cardiomyopathy
Acronym: BE STRONG HCM
Status: Completed | Type: Observational
Sponsor: Heartcenter, University Medical Center St. Radboud (Other)
Responsible Party: Principal Investigator, D.H.F. Gommans, MD, Principal Investigator, Heartcenter, University Medical Center St. Radboud
Other Study IDs: NL37776.091.11
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Troponin; Exercise; MRI
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Clinical HCM patients: Patients with an echocardiographically proven hypertrophic cardiomyopathy according to the ESC and ACCF/AHA guidelines
- Pre-clinical HCM patients: Individuals with a HCM associated mutation without the clinical characteristics of hypertrophic cardiomyopathy

SUMMARY:
Study population: 1) mutation carriers without the hypertrophic phenotype (pre-clinical Hypertrophic Cardiomyopathy (HCM)) and in 2) patients with clinically overt HCM (clinical HCM).

Hypothesis: Cardiac troponin release after exercise can be demonstrated in both clinical and pre-clinical HCM patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an echocardiographically proven hypertrophic cardiomyopathy according to the ESC guidelines or individuals with a HCM associated mutation without the clinical characteristics of hypertrophic cardiomyopathy (pre-clinical HCM patients);
* Age ≥ 18 years;
* Able to comply with the protocol;
* Written informed consent.

Exclusion Criteria:

* Known significant epicardial coronary artery disease;
* Patients with LVH in the clinical setting of other disorders that explain the myocardial hypertrophy (amyloidosis, MELAS, Anderson-Fabry, WPW etc.);
* Heart failure NYHA class III-IV;
* Patients with known hemodynamic instability or syncope during exercise due to left ventricular outflow gradient or occurrence of ventricular arrhythmia;
* History of PTSMA (percutaneous transluminal septal myocardial ablation) or Morrow myectomy;
* Patients not able to complete a bicycle test;
* Any contraindication to MR imaging (MR imaging is not obligatory for assessment of the primary objective, therefore relative exclusion criterion);
* Recent (within 30 days) admittance to the hospital for any cardiac reason (myocardial infarction, heart failure, cardiac arrhythmia, etc.);
* Severe renal insufficiency (eGFR < 30 ml/min);
* Any other condition which, in the opinion of the investigator, may pose a significant hazard to the subject if he or she participates in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of clinical or pre-clinical HCM patients that are registered in the HCM database of the HCM outpatient clinic of University Medical Center St. Radboud. This database will be screened for eligible patients according to the in- and exclusion criteria described below.
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Troponin levels at baseline and troponin rise after exercise testing using a high sensitivity-troponin (hs-troponin) assay | Baseline, 6 and 24 hours after exercise

SECONDARY OUTCOMES:
Correlation between troponin levels and phenotypic characteristics assessed with MRI (LV volumes, mass and ejection fraction, presence of LGE and/or elevated signal on T2-weighted imaging) | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Heartcenter, University Medical Center St. Radboud, Nijmegen, Gelderland, Netherlands